CLINICAL TRIAL: NCT01218763
Title: CANadian Clinical Evaluation of the Automatic Arrhythmia DETECTion in SpiderFlash™ Device
Brief Title: CANadian Clinical Evaluation of SpiderFlash Arrhythmia DETECTion in SpiderFlash™ Device
Acronym: CAN-DETECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sorin Group Canada (Industry)
Responsible Party: Marcio Sturmer, MD, Hopital du Sacre-Coeur, Montreal, Quebec
Other Study IDs: ITHO02
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2010-04

CONDITIONS: Arrhythmias, Cardiac
Keywords: Cardiac Event recorder; Sensitivity; Efficacy
MeSH Terms: conditions — Arrhythmias, Cardiac; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD patients: Candidates may come from the investigator's general population, who require DR ICD or CRT-D therapy for primary or secondary ICD indication and meet all study eligibility criteria

SUMMARY:
This clinical investigation is a prospective, non-randomized, multi-center pivotal trial.

This trial aims to validate the automatic detection features provided by the external long-duration SpiderFlash-t™ Event recorder coupled with its analyser EventScope™, and to assess the performances of the Mode Switch function provided by Sorin Group Implantable Cardioverter-Defibrillators (ICDs).

This trial is being performed first in order to demonstrate the ventricular tachycardia (VT)/ ventricular fibrillation (VF) sensitivity of the automatic VT/VF detection function of the EventScope™ software.

Patients will be implanted with an ICD from Sorin Group, with PARAD+ arrhythmia detection enabled and Mode Switch (MS) algorithms activated in all patients.

Arrhythmic events will be documented over a period of 6 to 8 weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

Patients already implanted with an OVATIO DR or CRT-D device may be included in the study if they presented with at least one clinical VT/VF event at the follow-up visit preceding the enrolment.

ICD or CRT-D device upgrading or replacement are allowed but under the condition that existing bipolar RV sensing/pacing lead and/or defibrillation lead and/or LV pacing lead (where applicable) are not of poor or questionable integrity.

Patients with implanted pacemakers may be included in the study only if the pacemaker is to be explanted or otherwise disabled prior to implanting the ICD or CRT-D system, to avoid any potential pacemaker-ICD interactions.

Patients must comply with all the following criteria in order to be included in the CAN-DETECT study:

1. Patient is eligible for implantation of a dual-chamber ICD or a CRT-D device according to current available guidelines for primary or secondary ICD indication .
2. A stable, optimal (as determined by the enrolling physician) drug regimen
3. Scheduled for implant of an OVATIO DR Model 6550 or OVATIO CRT 6750 or an equivalent device from Sorin Group.
4. Signed and dated informed consent.

Exclusion Criteria:

Any patient complying with any of the following criteria cannot be included in the CAN-DETECT study:

1. Any contraindication for standard cardiac pacing
2. Any contraindication for ICD therapy
3. Permanent high-degree AV Block for patients planned for dual-chamber ICD implant only.
4. Permanent AF for patients planned for dual-chamber ICD implant only.
5. Abdominal implantation site
6. Acute myocarditis
7. Mechanical tricuspid valve
8. Heart transplant recipient
9. Already participating in another clinical study
10. Life expectancy less than 6 months
11. Inability to understand the purpose of the study or refusal to cooperate
12. Inability or refusal to provide informed consent
13. Unavailability for scheduled follow-up at the implanting center
14. Under guardianship
15. Age of less than 18 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Candidates may come from the investigator's general population, who require DR ICD or CRT-D therapy for primary or secondary ICD indication and meet all study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2010-04

PRIMARY OUTCOMES:
VT/VF sensitivity | 2 years
  The primary purpose of this study is to evaluate the performance of the automatic detection of ventricular tachycardia and ventricular fibrillation (VT/VF) by the EventScope™ analyzer found in the Holter monitor SpiderFlash-t™. In order to validate this objective we will use the arrhythmia data collected in the memory storage found in the Sorin Group DR and CRT ICDs.

SECONDARY OUTCOMES:
AF sensitivity | 2 years
  The main secondary objective of this study is to evaluate the detection of atrial fibrillation by the Mode Switch algorithm found in the Sorin Group defibrillators. However, as SpiderFlash-t has only been validated on patients with spontaneous rhythm, in order to achieve this objective we will use the AF events detected by the EventScope™ in patients presenting with a spontaneous rhythm. SafeR mode, programmed in DR devices, will permit preservation of such rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Sturmer, MD, Principal Investigator — Hopital du Sacre-Coeur, Montreal, Qc, Canada; Bernard Thibault, MD, Principal Investigator — MHI, Montreal, Qc, Canada
Locations (5):
- Canada (5):
  - Grey-Nuns and Royal-Alexandra Hospitals, Edmonton, Alberta
  - Hotel-Dieu, Montreal, Quebec
  - Hopital du Sacre-Coeur, Montreal, Quebec
  - ICM, Montreal, Quebec
  - CHUS, Sherbrooke, Quebec